CLINICAL TRIAL: NCT04620863
Title: TRANSCRANIAL DIRECT CURRENT STIMULATION (t-DCS) AS ADD-ON TO NEUROREHABILITATION OF PISA SYNDROME IN PARKINSON DISEASE: A RANDOMIZED CONTROLLED TRIAL
Brief Title: TRANSCRANIAL DIRECT CURRENT STIMULATION (t-DCS) AS ADD-ON TO NEUROREHABILITATION OF PISA SYNDROME IN PARKINSON DISEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pisa-tDCS
Record Dates: First submitted 2020-10-26; First posted 2020-11-09 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-10

CONDITIONS: Parkinson Disease; Pisa Syndrome
Keywords: Parkinson Disease; Pisa Syndrome; Transcranial direct current stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Intervention Model Description: The study was a randomized, double-blind, controlled trial
Who Masked: Participant, Investigator
Masking Description: Transcranial direct current stimulation (t-DCS) was delivered by an expert technician (V.G.) that was not otherwise involved in the management of the patients. The managing physician as well as the physiotherapist were instead blind to the type of stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS group (Experimental): Patients randomized to the experimental group were treated with the following parameters: duration of stimulation of 20 minutes per session with a 2 mA intensity delivered at anodal and cathodal levels.
  Interventions: Other: t-DCS group
- Sham Group (Sham Comparator): The stimulation setting was exactly the same of the experimental group but the stimulation intensity was set according to a ramping up/ramping down method and delivered only in the first and last 30 seconds of each session. This stimulation paradigm is insufficient to produce a meaningful therapeutic effect, but it is necessary to guarantee the blind condition as it mimics the possible initial tingling sensation associated with active stimulation.
  Interventions: Other: Sham group

INTERVENTIONS:
Other: t-DCS group — All the participants received daily stimulation sessions for 5 consecutive days, starting from the first Monday after hospital admission (Monday to Friday). The primary motor cortex (M1) was identified using the International 10-20 system for C3 (left M1) or C4 (right M1). For the stimulation, the anode was placed over the primary motor cortex (M1) ipsilateral to the side of trunk deviation, and the cathode was placed over the primary motor cortex (M1) contralateral to the side of trunk deviation (bi-hemispheric stimulation).
  Arms: tDCS group
Other: Sham group — The stimulation setting was exactly the same but the stimulation intensity was set according to a ramping up/ramping down method and delivered only in the first and last 30 seconds of each session. This stimulation paradigm is insufficient to produce a meaningful therapeutic effect, but it is necessary to guarantee the blind condition as it mimics the possible initial tingling sensation associated with active stimulation.
  Arms: Sham Group

SUMMARY:
Pisa Syndrome (PS) is a lateral trunk flexion frequently associated to Parkinson's disease (PD). The management of PS is still a challenge for the clinician, because it poorly responds to anti-parkinsonian drugs, and the improvement achieved with neurorehabilitation or botulinum toxin injections tends to fade in 6 months or less. Transcranial direct current stimulation (t-DCS) is a non-invasive neuromodulation technique, with promising results in movement disorders. Aim of our study is to evaluate the role of bi-hemispheric t-DCS as add-on to neurorehabilitation in PS. Twenty-eight patients affected by PD and PS were managed with a 4-week hospital neurorehabilitation programme and randomized to: 1) t-DCS group: 5 daily sessions (20 minutes - 2 mA) with cathode over the primary motor cortex (M1) contralateral to PS, and anode over the M1 cortex ipsilateral to PS; or 2) sham group. Patients were tested with kinematic analysis of trunk movement in static and dynamic conditions, UPDRS-III, FIM, and VAS for lumbar pain rating at hospital admission (T0), at hospital discharge (end of neurorehabilitation - T1), and 6 months later (T2). At T0, the evaluations were completed by an EMG study of trunk muscles activation.

DETAILED DESCRIPTION:
Axial disorders are frequent complications of Parkinson's Disease (PD) and they can lead to postural deformities and balance impairments. The most prevalent postural disorders of PD are represented by camptocormia, antecollis, scoliosis, and Pisa syndrome (PS).

The pathogenesis of these disorders has not yet been completely elucidated, and it is characterized by a complex interlacement between central and peripheral mechanisms.

The first report of PS dates back in 1972, when Ekobm described a case series of three patients who developed a lateral trunk flexion in close temporal relationship with neuroleptics assumption. The roster of drugs associated with an acute/subacute onset of PS is huge and constantly growing, and it includes: antidepressants (mirtazapine, sertraline), cholinesterase inhibitor (rivastigmine, galantamine, donepezil), neuroleptics (tiapride, clotiapine, clozapine, aipiprazole, butyrophenone, paliperidone, quetiapine), dopamine agonists, (pramipexolo, ropinirole, pergolide), lithium, valproic acid, and betahistine. Nonetheless, PS was described as well in patients with neurodegenerative disorders, and in particular in PD and parkinsonism without drugs exposure.

The prevalence of PS is around 8.3% (9.3% in women and 6.4% in men) when calculated in a psychogeriatric population, and it is 8 to 8.8% when populations of PD patients were considered.

Formal diagnostic criteria for PS are not available, indeed the diagnosis is based on the clinical features:

* presence of a lateral flexion of the trunk with a homogenous angle between sacrum and spinous process of the 7th cervical vertebra;
* association of an ipsilateral rotation of the trunk around the sagittal axis that leads to a higher and anterior position of the shoulder contralateral to the side of trunk deviation;
* the postural disorder worsens during standing position, sitting position and gait;
* the postural disorder improves in supine position;
* disregard of patients for the postural disorder.

The fluctuation of the postural alteration during static (supine position vs. upright standing position) and dynamic conditions appears to be crucial to differentiate PS from scoliosis.

A lateral trunk deviation of at least 10° is commonly accepted for the diagnosis, although higher or lower cut-offs were used in the past. According to the degree of the lateral trunk flexion, PS can be further divided in mild (less than 20°) or severe (more than 20°) phenotypes.

Patients with PD and PS showed some typical clinical and demographic features when compared to PD patients without postural alterations: they are older, PD is longer in duration, more severe and with a more pronounced asymmetry of motor symptoms. The parkinsonian symptoms involving the upper limbs as well as gait impairment are more severe in PD patients with PS. Moreover, they are characterized by a higher incidence of falls, arthrosis, osteoporosis, orthopedics diseases and pain, specifically lumbar and lower back pain, which is reported in up to 75% of patients with PD and PS.

The management of PS is still a challenge for the physician. PS poorly responds to antiparkinsonian drugs, although there aren't studies specifically designed to assess this topic.

Neurorehabilitation represents one of the fundamental approach to PD and to postural disorders in general, not only for the treatment of the motor symptoms itself but also to improve quality of life and autonomy in the activity of daily living.

The study was a randomized, double-blind, controlled trial aimed to assess the efficacy of five daily sessions of bi-hemispheric t-DCS in add-on to an in-hospital neurorehabilitation protocol in patients affected by PD and PS.

At hospital admission (T0 - baseline), all patients underwent complete neurological, general and functional examinations by a Neurologist with expertise in movement disorders and neurorehabilitation. Patients who fulfilled inclusion and exclusion criteria underwent a baseline kinematic analysis of trunk movement. Patients with at least 10° of lateral trunk flexion completed the baseline evaluations with a dynamic electromyographic (EMG) study of trunk muscles, and with administration of a set clinical scales for the evaluations of motor disability, functional independence, and lumbar pain.

After that, patients were randomly assigned to "t-DCS" or "sham" treatment, and they started the double-blind phase of the study. The 5-day t-DCS/sham treatment was delivered in 5 daily consecutive sessions, starting from the first Monday after hospital admission. In parallel to neuromodulation, all patients were treated with a standardized 4-week rehabilitation programme. The kinematic analysis of trunk movement as well as the administration of the set of questionnaires were repeated at the end of the 4-week rehabilitation programme (T1 - hospital discharge), and 6 months after discharge (T2).

The randomization was performed according to a block randomization method. A unique randomization list was generated before enrollment with the following parameters: 6 blocks; 6 patients per block (3 for t-DCS group, and 3 for sham group).

All the patients were treated with an optimized and individualized anti-parkinsonian therapy, which dose and regimen were kept stable during the overall study period. All the evaluations were performed in the morning, and always in an ON phase.

The specific and standardized in-hospital rehabilitation programme was focused on the rehabilitation of the trunk postural disorder. All patients were treated with 90-minute daily sessions, 6 days a week (Monday to Saturday) for four weeks.

Each session was structured as follow:

* 10 minutes of cardiovascular warm-up activities: intersegmental coordination exercises; exercises to release shoulder and pelvic girdle; pelvic anteversion and retroversion movements to improve diaphragmatic respiration (supine position); breathing exercises to promote expansion of the chest;
* 15 minutes of stretching exercises: exercises to stretch the muscles of the posterior kinematic chain; exercises to stretch the pectoralis muscles; exercises to stretch the ischio-cruralis muscles; assumption of the prone position, sitting on heels and stretching the arms out in front; the "bridge" exercise to stretch the muscles of the anterior abdominal wall, glutei, quadriceps and hamstring; exercises to stretch lumbar muscles (in the supine position, each knee, in turn, is brought to the chest);
* 15 minutes of strengthening exercises in a functional context: exercises to strengthen the dorsal muscles (arms extended and hands outstretched as though to take something); lateral bending (arms lying along the body and hands reaching down as though to pick up something); stretching using the wall bars;
* 20 minutes of gait training: overground gait training (forwards, backwards, and lateral); walking on the spot;
* 15 minutes of balance training: path with obstacles; balance exercises performed in order of difficulty (heel-to-toe walking, lateral walking crossing the legs, walking along a path on surfaces of different texture);
* 15 minutes of relaxation exercises: intersegmental coordination exercises; segmental passive mobilization (until maximum joint range of motion is reached); breathing exercises to promote expansion of the chest.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years;
* Hoehn and Yahr stage between II and III;
* Mini-Mental State Examination score above 24;
* lateral trunk flexion of at least 10° at baseline.

Exclusion Criteria:

* history of major psychiatric or other neurological conditions;
* history of back surgery, tumors or infections of the spine, intradural or extradural hematoma, ankylosing spondylitis, spinal stenosis;
* history of idiopathic scoliosis;
* botulin toxin treatment in the previous year;
* any change in dose or regimen of the anti-parkinsonian therapy in the last month before enrolment.

Thirty patients affected by Parkinson' Disease (PD) and Pisa Syndrome (PS) were consecutive enrolled among those attending the Neurorehabilitation Department of the IRCCS Mondino Foundation (Pavia, Italy). Idiopathic PD was diagnosed according to the Movement Disorders Society clinical diagnostic criteria for PD. Pisa syndrome was clinically diagnosed according to the following criteria:

* a lateral flexion of the trunk with a homogenous angle between sacrum and spinous process of the 7th cervical vertebra;
* an ipsilateral axial rotation of the trunk around the sagittal axis, that leads to a higher and anterior position of the shoulder contralateral to the side of trunk deviation;
* the worsening of the postural disorder during standing position, sitting position and gait;
* the improvement of the postural disorder in supine position.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
Change of Stat Tot (Stat Bend + Stat Flex) | Change from Baseline at 28 weeks (T2)
  Total postural alteration in the upright standing position (Stat Tot): lateral trunk inclination in the upright standing position (Stat Bend) plus anterior trunk flexion in the upright standing position (Stat Flex).

SECONDARY OUTCOMES:
Change of Stat Bend | Change from Baseline at 28 weeks (T2)
  Lateral trunk inclination in the upright standing position
Change of Stat Flex | Change from Baseline at 28 weeks (T2)
  Anterior trunk flexion in the upright standing position
Change of ROM Ips | Change from Baseline at 28 weeks (T2)
  Range of Motion (ROM) of trunk bending ipsilateral to the side of trunk deviation
Change of ROM Con | Change from Baseline at 28 weeks (T2)
  Range of Motion (ROM) of trunk bending contralateral to the side of trunk deviation
Change of ROM flex | Change from Baseline at 28 weeks (T2)
  Range of Motion (ROM) of anterior trunk flexion
Change of ROM Ext | Change from Baseline at 28 weeks (T2)
  Range of Motion (ROM) of posterior trunk extension
Change of Total ROM of the trunk | Change from Baseline at 28 weeks (T2)
  ROM Ips + ROM Con + ROM Flex + ROM Ext
Change of The Unified Parkinson's Disease Rating Scale - part III - Motor examination (UPDRS-III) | Change from Baseline at 28 weeks (T2)
  It consists of 18 items (score from 0 to 4). Higher scores are worst otcomes.
Change of Functional Independence Measure (FIM) | Change from Baseline at 28 weeks (T2)
  The Functional Independence Measure (FIM) is an 18-item measurement tool that explores an individual's physical, psychological and social function. FIM scores range from 1 to 7 (1= total assist and 7= complete independence).
Change of Visual analog scale (VAS). | Change from Baseline at 28 weeks (T2)
  Lumbar pain severity was rated according to a 0 to 10 visual analog scale. Zero is no pain and 10 is worst pain.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Tassorelli, MD, Study Director — IRCCS Mondino Foundation, Pavia
Locations (1):
- Neurorehabilitation Department, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ekbom K, Lindholm H, Ljungberg L. New dystonic syndrome associated with butyrophenone therapy. Z Neurol. 1972;202(2):94-103. doi: 10.1007/BF00316159. No abstract available. PMID 4115928
- [Background] Gambarin M, Antonini A, Moretto G, Bovi P, Romito S, Fiaschi A, Tinazzi M. Pisa syndrome without neuroleptic exposure in a patient with Parkinson's disease: case report. Mov Disord. 2006 Feb;21(2):270-3. doi: 10.1002/mds.20711. PMID 16161148
- [Background] Barone P, Santangelo G, Amboni M, Pellecchia MT, Vitale C. Pisa syndrome in Parkinson's disease and parkinsonism: clinical features, pathophysiology, and treatment. Lancet Neurol. 2016 Sep;15(10):1063-74. doi: 10.1016/S1474-4422(16)30173-9. Epub 2016 Aug 8. PMID 27571158
- [Background] Tinazzi M, Gandolfi M, Ceravolo R, Capecci M, Andrenelli E, Ceravolo MG, Bonanni L, Onofrj M, Vitale M, Catalan M, Polverino P, Bertolotti C, Mazzucchi S, Giannoni S, Smania N, Tamburin S, Vacca L, Stocchi F, Radicati FG, Artusi CA, Zibetti M, Lopiano L, Fasano A, Geroin C. Postural Abnormalities in Parkinson's Disease: An Epidemiological and Clinical Multicenter Study. Mov Disord Clin Pract. 2019 Jun 29;6(7):576-585. doi: 10.1002/mdc3.12810. eCollection 2019 Sep. PMID 31538092
- [Background] Tinazzi M, Fasano A, Geroin C, Morgante F, Ceravolo R, Rossi S, Thomas A, Fabbrini G, Bentivoglio A, Tamma F, Cossu G, Modugno N, Zappia M, Volonte MA, Dallocchio C, Abbruzzese G, Pacchetti C, Marconi R, Defazio G, Canesi M, Cannas A, Pisani A, Mirandola R, Barone P, Vitale C; Italian Pisa Syndrome Study Group. Pisa syndrome in Parkinson disease: An observational multicenter Italian study. Neurology. 2015 Nov 17;85(20):1769-79. doi: 10.1212/WNL.0000000000002122. Epub 2015 Oct 21. PMID 26491088
- [Background] Tassorelli C, Furnari A, Buscone S, Alfonsi E, Pacchetti C, Zangaglia R, Pichiecchio A, Bastianello S, Lozza A, Allena M, Bolla M, Sandrini G, Nappi G, Martignoni E. Pisa syndrome in Parkinson's disease: clinical, electromyographic, and radiological characterization. Mov Disord. 2012 Feb;27(2):227-35. doi: 10.1002/mds.23930. Epub 2011 Oct 13. PMID 21997192
- [Background] Doherty KM, Davagnanam I, Molloy S, Silveira-Moriyama L, Lees AJ. Pisa syndrome in Parkinson's disease: a mobile or fixed deformity? J Neurol Neurosurg Psychiatry. 2013 Dec;84(12):1400-3. doi: 10.1136/jnnp-2012-304700. Epub 2013 Mar 26. PMID 23532719
- [Background] Bonanni L, Thomas A, Varanese S, Scorrano V, Onofrj M. Botulinum toxin treatment of lateral axial dystonia in Parkinsonism. Mov Disord. 2007 Oct 31;22(14):2097-103. doi: 10.1002/mds.21694. PMID 17685467
- [Background] Etoom M, Alwardat M, Aburub AS, Lena F, Fabbrizo R, Modugno N, Centonze D. Therapeutic interventions for Pisa syndrome in idiopathic Parkinson's disease. A Scoping Systematic Review. Clin Neurol Neurosurg. 2020 Nov;198:106242. doi: 10.1016/j.clineuro.2020.106242. Epub 2020 Sep 18. PMID 32979681
- [Background] Tinazzi M, Geroin C, Gandolfi M, Smania N, Tamburin S, Morgante F, Fasano A. Pisa syndrome in Parkinson's disease: An integrated approach from pathophysiology to management. Mov Disord. 2016 Dec;31(12):1785-1795. doi: 10.1002/mds.26829. Epub 2016 Oct 25. PMID 27779784
- [Background] Tassorelli C, De Icco R, Alfonsi E, Bartolo M, Serrao M, Avenali M, De Paoli I, Conte C, Pozzi NG, Bramanti P, Nappi G, Sandrini G. Botulinum toxin type A potentiates the effect of neuromotor rehabilitation of Pisa syndrome in Parkinson disease: a placebo controlled study. Parkinsonism Relat Disord. 2014 Nov;20(11):1140-4. doi: 10.1016/j.parkreldis.2014.07.015. Epub 2014 Aug 13. PMID 25175601
- [Background] Castrioto A, Piscicelli C, Perennou D, Krack P, Debu B. The pathogenesis of Pisa syndrome in Parkinson's disease. Mov Disord. 2014 Aug;29(9):1100-7. doi: 10.1002/mds.25925. Epub 2014 Jun 7. PMID 24909134
- [Background] Di Matteo A, Fasano A, Squintani G, Ricciardi L, Bovi T, Fiaschi A, Barone P, Tinazzi M. Lateral trunk flexion in Parkinson's disease: EMG features disclose two different underlying pathophysiological mechanisms. J Neurol. 2011 May;258(5):740-5. doi: 10.1007/s00415-010-5822-y. Epub 2010 Nov 16. PMID 21079986
- [Background] Tinazzi M, Juergenson I, Squintani G, Vattemi G, Montemezzi S, Censi D, Barone P, Bovi T, Fasano A. Pisa syndrome in Parkinson's disease: an electrophysiological and imaging study. J Neurol. 2013 Aug;260(8):2138-48. doi: 10.1007/s00415-013-6945-8. Epub 2013 May 22. PMID 23695587
- [Background] Bartolo M, Serrao M, Tassorelli C, Don R, Ranavolo A, Draicchio F, Pacchetti C, Buscone S, Perrotta A, Furnari A, Bramanti P, Padua L, Pierelli F, Sandrini G. Four-week trunk-specific rehabilitation treatment improves lateral trunk flexion in Parkinson's disease. Mov Disord. 2010 Feb 15;25(3):325-31. doi: 10.1002/mds.23007. PMID 20131386
- [Background] Nitsche MA, Liebetanz D, Antal A, Lang N, Tergau F, Paulus W. Modulation of cortical excitability by weak direct current stimulation--technical, safety and functional aspects. Suppl Clin Neurophysiol. 2003;56:255-76. doi: 10.1016/s1567-424x(09)70230-2. No abstract available. PMID 14677403
- [Background] DaSilva AF, Volz MS, Bikson M, Fregni F. Electrode positioning and montage in transcranial direct current stimulation. J Vis Exp. 2011 May 23;(51):2744. doi: 10.3791/2744. PMID 21654618
- [Background] Lefaucheur JP, Andre-Obadia N, Antal A, Ayache SS, Baeken C, Benninger DH, Cantello RM, Cincotta M, de Carvalho M, De Ridder D, Devanne H, Di Lazzaro V, Filipovic SR, Hummel FC, Jaaskelainen SK, Kimiskidis VK, Koch G, Langguth B, Nyffeler T, Oliviero A, Padberg F, Poulet E, Rossi S, Rossini PM, Rothwell JC, Schonfeldt-Lecuona C, Siebner HR, Slotema CW, Stagg CJ, Valls-Sole J, Ziemann U, Paulus W, Garcia-Larrea L. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS). Clin Neurophysiol. 2014 Nov;125(11):2150-2206. doi: 10.1016/j.clinph.2014.05.021. Epub 2014 Jun 5. PMID 25034472
- [Result] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for idiopathic Parkinson's disease. Cochrane Database Syst Rev. 2016 Jul 18;7(7):CD010916. doi: 10.1002/14651858.CD010916.pub2. PMID 27425786